CLINICAL TRIAL: NCT01848769
Title: A Single-dose, Open-Label, 2-Way Cross-Over, Clinical Pharmacology Study Of Chf 1535 50/6 HFA pMDI (Fixed Combination Of Beclomethasone Dipropionate 50µg Plus Formoterol Fumarate 6 µg) Using The Aerochamber Plus™ Spacer Device Versus The Free Combination Of Beclomethasone HFA pMDI And Formoterol HFA pMDI Available On The Market Using The Aerochamber Plus™ Spacer Device In Asthmatic Children
Brief Title: Clinical Pharmacology Study of CHF1535 pMDI 50/6 µg Versus The Free Combination In Asthmatic Children 5-11 Years Old
Acronym: PAED1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-0902-PR-0013
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Asthma
Keywords: Asthma; ICS+LABA; Children; Inhalation; pMDI
MeSH Terms: conditions — Asthma; Respiratory Aspiration | interventions — alpha-ketoisovalerate dehydrogenase phosphatase; Beclomethasone; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF1535 pMDI + AC Plus (Experimental): Fixed combination of Beclomethasone Dipropionate and Formoterol 50/6 mcg with Aerochamber Plus spacer device
  Interventions: Drug: CHF1535 pMDI + AC Plus
- BDP and Formoterol + AC Plus (Active Comparator): Beclomethasone Dipropionate 50 mcg and Formoterol 6 mcg with Aerochamber Plus spacer device
  Interventions: Drug: BDP + AC Plus; Drug: Formoterol + AC Plus

INTERVENTIONS:
Drug: CHF1535 pMDI + AC Plus — Four inhalations for a total dose of BDP/FF 200/24 mcg
  Other Names: Fixed combination of BDP and FF 50/6 mcg
  Arms: CHF1535 pMDI + AC Plus
Drug: BDP + AC Plus — Four inhalations for a total dose of BDP 200 mcg
  Other Names: Beclomethasone Dipropionate 50 mcg with Aerochamber Plus
  Arms: BDP and Formoterol + AC Plus
Drug: Formoterol + AC Plus — Four inhalations for a total dose of Formoterol 24 mcg
  Other Names: Formoterol 6 mcg with Aerochamebr Plus
  Arms: BDP and Formoterol + AC Plus

SUMMARY:
The rationale is to investigate the systemic availability of BDP/B17MP and formoterol after single oral inhalation of CHF 1535 50/6 pMDI vs the free combination of approved BDP and Formoterol pMDIs, in asthmatic children (5 to 11 years old).

ELIGIBILITY:
Inclusion Criteria:

* Male/Female children aged 5-11 years
* Written informed consent obtained by parents/legal representative (according to local regulation) and by the minor (age and local regulation permitting).
* children with stable asthma on regular treatment with ICS or using short-acting inhaled beta2-agonists as reliever to control asthma symptoms
* Forced expiratory volume in one second (FEV1) > 70% of predicted values (% pred) after withholding beta2-agonist treatment for a minimum of 4 h prior to each dose period.

  6. A cooperative attitude and ability to be trained about the proper use of pMDI with a spacer device and compliant to study procedures.

Exclusion Criteria:

* Past or present diagnoses of cardiovascular, renal or liver disease
* Known hypersensitivity to the active treatments
* Exacerbation of asthma symptoms within the previous 4 weeks
* Inability to perform the required breathing technique and blood sampling
* Hospitalization due to exacerbation of asthma within 1 month prior to inclusion
* Lower respiratory tract infection within 1 month prior to inclusion
* Disease (other than asthma) which might influence the outcome of the study
* Obesity, i.e. > 97% weight percentile by local standards

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
B17MP AUC0-t | pre-dose until 8hours post dose
  B17MP (active metabolite of BDP) systemic exposure as AUC0-t

SECONDARY OUTCOMES:
B17MP PK profile | pre-dose until 8 hours post-dose
BDP PK prolile | Pre-dose until 8 hours post-dose
Formoterol PK profile | Pre-dose until 8 hours post-dose
Plasma potassium AUC, Cmin, tmin | Pre-dose until 8 hours post-dose
  Plasma potassium to evaluate drug systemic effect
Urinary Cortisol excretion | Pre-dose until 8 hours post-dose
  8h urinary excretion of cortisol and 8h urinary excretion of cortisol normalized for 8h creatinine excretion to evaluate dru systemic effects
Glucose in urine | Pre-dose until 8 hours post-dose
  Glucose to evaluate the drug systemic effects
Heart rate Time averaged heart rate value (AUC0-t)/t | Pre-dose until 8 hours post-dose
  Heart rate to evaluate the drug systemic effects
Spirometry: PEF | Pre-dose until 8 hours post-dose
  Peak respiratory flow as a measure of drug efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Hans Bisgaard, MD DMSci, Principal Investigator — BorneAstmaKlinikken
Locations (1):
- BorneAstmaKlinikken, Copenhagen, Denmark

REFERENCES:
- [Background] Govoni M, Piccinno A, Lucci G, Poli G, Acerbi D, Baronio R, Singh D, Kuna P, Chawes BL, Bisgaard H. The systemic exposure to inhaled beclometasone/formoterol pMDI with valved holding chamber is independent of age and body size. Pulm Pharmacol Ther. 2015 Feb;30:102-9. doi: 10.1016/j.pupt.2014.04.003. Epub 2014 Apr 16. PMID 24746942
- [Result] Chawes BL, Piccinno A, Kreiner-Moller E, Vissing NH, Poorisrisak P, Mortensen L, Nilson E, Bisgaard A, Dossing A, Deleuran M, Skytt NL, Samandari N, Sergio F, Ciurlia G, Poli G, Acerbi D, Bisgaard H. Pharmacokinetic comparison of inhaled fixed combination vs. the free combination of beclomethasone and formoterol pMDIs in asthmatic children. Br J Clin Pharmacol. 2013 Apr;75(4):1081-8. doi: 10.1111/j.1365-2125.2012.04459.x. PMID 22978252
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2009-010434-22